CLINICAL TRIAL: NCT03001583
Title: Clinical Trial Comparing Two Health Education Programs for Obese Patients: Groups With Health Education Plus Cooking Program vs. Only Education Without Cooking
Brief Title: Clinical Trial Comparing Two Health Education Programs for Obese Patients (HEPO-TRIAL)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators hadn't got funding to support the study
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRUCO_2016
Record Dates: First submitted 2016-12-07; First posted 2016-12-23 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: Mediterranean diet; weight loss; type 2 diabetes; education program; cooking
MeSH Terms: conditions — Obesity; Weight Loss; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Program with cooking lessons (Experimental): Structured education program of mediterranean diet and lifestyle changes with cooking lessons delivered in monthly visits for an induction phase of 6 months, with an extension period of up to two years.
  Interventions: Behavioral: Education program with cooking lessons
- Education without cooking (Active Comparator): Structured education program of mediterranean diet and lifestyle changes WITHOUT cooking lessons delivered in monthly visits for an induction phase of 6 months, with an extension period of up to two years.
  Interventions: Behavioral: Education program WITHOUT cooking lessons

INTERVENTIONS:
Behavioral: Education program with cooking lessons — Structured education program of mediterranean diet and lifestyle changes with cooking lessons delivered in monthly visits for an induction phase of 6 months, with an extension period of up to two years.
  Arms: Education Program with cooking lessons
Behavioral: Education program WITHOUT cooking lessons — Structured education program of mediterranean diet and lifestyle changes WITHOUT cooking lessons delivered in monthly visits for an induction phase of 6 months, with an extension period of up to two years.
  Arms: Education without cooking

SUMMARY:
Clinical trial comparing two health education programs for obese patients in order to achieve a substantial and beneficial weight loss, using mediterranean diet. Patients will be allocated to two groups, one will receive education in diet and lifestyle, and the other one the same plus cooking lessons. The intervention period is for 6 months with monthly visits and phone and email contacts in between. An extension observation period of two years is also planned with 6 months contacts in our clinic, also with phone and email contact available.

DETAILED DESCRIPTION:
Eligibility: obese patients attending our center. Exclusion criteria: previous dietary or anti-obesity drugs treatments, previous bariatric surgery, eating disorders, desire for short-term bariatric surgery, active neoplasia, end stage kidney or liver disease, food allergies or celiac disease.

Sample Size: a total of 260 patients (130 patients in each group) are needed for α=0.05 and 1-ß=0.8, to reach a difference of a 5% in weight loss between both groups, with a maximum of a 30% dropouts.

Intervention: structured health education program of Mediterranean diet and lifestyle changes with cooking lessons in monthly sessions, with the aid of phone and email contacts during an induction phase of 6 months, followed by an extension period of 18 months.

Control: same strategy without the cooking lessons. Primary outcome: weight loss in % Secondary outcomes: reversal in obesity associated comorbidities and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients attending our center

Exclusion Criteria:

* Previous dietary or pharmacologic treatment for obesity, previous bariatric surgery, desired bariatric surgery in the short-term, eating disorders, end-stage kidney or liver disease, active neoplasia, food allergies, celiac disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 6 months

SECONDARY OUTCOMES:
Weight loss | Visits at 12, 18 and 24 months (to complete a total study time period of 24 months)